CLINICAL TRIAL: NCT00515528
Title: Randomized Phase II Study of Multipeptide Vaccination With or Without Regulatory T Cell Depletion Using Ontak in Patients With Metastatic Melanoma
Brief Title: Vaccination Plus Ontak in Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The immune monitoring data failed to demonstrate an improvement in any biologic endpoint with denileukin diftitox.
Sponsor: University of Chicago (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15232B
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Melanoma
Keywords: metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine Alone (Experimental): Subjects received vaccine immunization injected intra-dermally or subcutaneously on day 1. The vaccine was an emulsification consisting of 250 mcg each of the following peptides: Melan-A, gp100, MAGE-3, and NA17 as well as GM-CSF 125 mcg and Montanide. A second and third vaccination was given at 2 weeks and 4 weeks after the first. If there was no evidence of cancer progression, additional courses of three vaccinations administered at 2 week intervals were administered until disease progression.
  Interventions: Biological: 4-peptide melanoma vaccine
- Vaccine plus Ontak (Experimental): Subjects in Vaccine plus Ontak received the same vaccination strategy as Vaccine alone group but additionally received a single dose of denileukin diftitox(18 mcg/kg) 4 days prior to the first vaccine administration
  Interventions: Biological: 4-peptide melanoma vaccine; Drug: Ontak

INTERVENTIONS:
Biological: 4-peptide melanoma vaccine — Experimental cancer vaccine given as a shot under the skin once every two weeks
Drug: Ontak — A single dose of Ontak given as an intravenous infusion over 30 minutes, 4 days before the first vaccine is given.
  Arms: Vaccine plus Ontak

SUMMARY:
The purpose of this study is to determine if an experimental melanoma vaccine can produce an immune response in patients with metastatic melanoma, and if combining this vaccine with the drug Ontak can improve these immune responses. It is also hoped that this will lead to tumor shrinkage.

DETAILED DESCRIPTION:
This is an open-label, randomized phase II, single institution study comparing administration of a 4-peptide melanoma vaccine alone or post-Ontak, in patients with metastatic melanoma.

Treatment:

1. Cohort A: Vaccine alone. Patients will receive immunization with an emulsion of 4 melanoma peptides (250 mcg each)/GM-CSF/Montanide injected intradermally/subcutaneously on day 1. A second vaccination will be given 2 weeks later and a third vaccination 2 weeks after that. Patients will be re-evaluated around week 6 and can continue courses of 3 vaccinations (one every 2 weeks) until disease progression.
2. Cohort B: Ontak plus vaccine. Patients will receive Ontak (18 mcg/kg) intravenously on day -4 for one dose. On day 0, they will receive the first immunization with an emulsion of 4 melanoma peptides (250 mcg each)/GM-CSF/Montanide injected intradermally/subcutaneously. A second vaccination will be given 2 weeks later and a third vaccination 2 weeks after that. Patients will be re-evaluated around week 6 and can continue courses of 3 vaccinations (one every 2 weeks) until disease progression. However, no further Ontak will be given.

Duration: Patients may remain on study until disease progression, unacceptable toxicity, patient choice to withdraw, or physician decision to discontinue therapy (due to intervening illness, poor patient compliance, or other situation that would increase patient risk).

ELIGIBILITY:
Inclusion Criteria:

* Melanoma with evidence of metastatic disease
* Life expectancy of at least 12 weeks.
* Karnofsky performance status index of greater than or equal to 80%.
* Adequate hematopoietic, renal, and hepatic function, defined as:
* Patient must express HLA-A2
* Tumor biopsy: patient must agree to undergo biopsy of accessible tumor before and after therapy, when feasible, to study tumor cell properties and characteristics of immune cells.
* EKG without evidence of arrhythmia or changes that indicate acute ischemia.
* Pulse oximetry showing oxygen saturation of at least 90% on room air.

Exclusion Criteria:

* Significant cardiovascular disease, or cardiac arrhythmia requiring medical intervention.
* Pregnant or nursing women.
* Biological therapy in the 4 weeks prior to the start of dosing.
* Patients with intrinsic immunosuppression, including seropositivity for HIV antibody.
* Serious concurrent infection, including active tuberculosis, hepatitis B, or hepatitis C.
* Concurrent systemic corticosteroids (except physiologic replacement doses)or other immunosuppressive drugs (eg. cyclosporin A).
* Psychiatric illness that may make compliance to the clinical protocol unmanageable or may compromise the ability of the patient to give informed consent.
* Active or history of autoimmune disease
* Active gastrointestinal bleeding or uncontrolled peptic ulcer disease.
* Presence of untreated brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-04-23 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gajeweski, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Luke JJ, Zha Y, Matijevich K, Gajewski TF. Single dose denileukin diftitox does not enhance vaccine-induced T cell responses or effectively deplete Tregs in advanced melanoma: immune monitoring and clinical results of a randomized phase II trial. J Immunother Cancer. 2016 Jun 21;4:35. doi: 10.1186/s40425-016-0140-2. eCollection 2016. PMID 27330808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine Alone | Vaccine Plus Ontak
Started | 10 | 7
Completed | 10 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine Alone | Vaccine Plus Ontak | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Median (Full Range); unit: years] | 57 [46 to 81] | 63 [45 to 77] | 63 [45 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Outcome
Description: Proportion of Patients With a Best Response of Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD).
  Response was evaluated every 6 weeks based on Response Evaluation In Solid Tumor (RECIST) version 1.1.
  Per RECIST v1.1 for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (PD); PD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Alone | Vaccine Plus Ontak
Number analyzed (Participants) | 10 | 7
Participants
  PR | 1 | 0
  SD | 4 | 4
  PD | 5 | 3

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Vaccine Alone | Vaccine Plus Ontak
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/7
Serious Adverse Events (participants affected / at risk) | 2/10 | 2/7
Other Adverse Events (participants affected / at risk) | 10/10 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Alone (N=10) | Vaccine Plus Ontak (N=7)
Syncope (Nervous system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pericardial tamponade (Congenital, familial and genetic disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine Alone (N=10) | Vaccine Plus Ontak (N=7)
Injection Site Pain (General disorders) | 7 | 3
Headache (General disorders) | 9 | 2
Fatigue (General disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Fever (General disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Infection (Infections and infestations) | 0 | 1
Respiratory (Respiratory, thoracic and mediastinal disorders) | 4 | 4
SGOT (Investigations) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
SGPT (Investigations) | 3 | 3
Anemia (Blood and lymphatic system disorders) | 1 | 1
Chills (General disorders) | 2 | 1
Absolute Neutrophil Count Decrease (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Insomnia (General disorders) | 1 | 0
Creatinine Increased (Investigations) | 2 | 1
Bilirubin increased (Investigations) | 2 | 0
Neurological (Nervous system disorders) | 3 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Visual Problems (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Neck Tightness (General disorders) | 1 | 0
Edema (Nervous system disorders) | 0 | 1
Weight Gain (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No